CLINICAL TRIAL: NCT02593448
Title: Influence of Cardiopulmonary Bypass and Sevoflurane or Propofol Anesthesia on Tissue Oxygen Saturation of Thenar Muscle in Adults.
Brief Title: Influence of Cardiopulmonary Bypass, and Sevoflurane or Propofol Anesthesia, on Tissue Oxygen Saturation.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Principal Investigator, Maciej M. Kowalik, Dr hab. med. Romuald Lango, Medical University of Gdansk
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NKBN/34/2012
Record Dates: First submitted 2015-10-27; First posted 2015-11-02 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-10

CONDITIONS: NIR Spectroscopy
Keywords: Cardiopulmonary Bypass; Anoxia
MeSH Terms: conditions — Hypoxia | interventions — Anesthesia, General

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Propofol (Active Comparator): General anaesthesia with Propofol use. Maintenance of anaesthesia in group P will be accomplished using continuous intravenous infusion of propofol 2-4 mg kg/h.
  Propofol infusion rate will be adjusted according to patient's haemodynamic parameters and the level of anaesthesia, as assessed with Bispectral Index (BIS), with a target range of 40-60.
  Intervention: NIRS during VOT on several timepoints.
  Interventions: Procedure: NIRS during VOT; Procedure: General anaesthesia with propofol use
- Sevoflurane (Experimental): General anaesthesia with sevoflurane use. Sevoflurane concentration in exhaled gas will be adjusted according to patient's haemodynamic parameters and the level of anaesthesia, as assessed with BIS, with a target range of 40-60.
  Intervention: NIRS during VOT on several timepoints.
  Interventions: Procedure: NIRS during VOT; Procedure: General anaesthesia with sevoflurane use

INTERVENTIONS:
Procedure: NIRS during VOT — Near infrared spectroscopy with INVOS oximeter during vascular occlusion test (VOT) on following timepoints:
  1. 30 minutes after anaesthesia induction,
  2. directly after the sternotomy,
  3. during CPB - 20 minutes after aortic cross-clamping ,
  4. 40 minutes after aortic cross-clamping,
  5. 20 minutes after the release of the aortic cross-clamp,
  6. 45 minutes after weaning of CPB.
Procedure: General anaesthesia with propofol use — Premedication: lorazepam 50 μg kg-1, omeprazole 40 mg, and metoprolol 12.5 mg one hour before transport to the operating theatre.
  Anaesthesia induction: 0.2 mg fentanyl, 0.3 mg/kg, etomidate, and vecuronium bromide 0.1 mg/kg for muscle relaxation, followed by a continuous infusion at the rate of 0.05 mg/kg/h until the sternum closure.
  Intraoperative analgesia: fentanyl in fractions, up to the total dose of 20-30 μg/kg.
  Maintenance of anaesthesia in 'Propofol' group will be accomplished using continuous intravenous infusion of propofol 2-4 mg kg/h.
  Propofol infusion rate will be adjusted according to patient's haemodynamic parameters and the level of anaesthesia, as assessed with Bispectral Index (BIS), with a target range of 40-60.
  Other Names: Propofol Total Intravenous Anesthesia (TIVA)
  Arms: Propofol
Procedure: General anaesthesia with sevoflurane use — Premedication: lorazepam 50 μg kg-1, omeprazole 40 mg, and metoprolol 12.5 mg one hour before transport to the operating theatre.
  Anaesthesia induction: 0.2 mg fentanyl, 0.3 mg/kg, etomidate, and vecuronium bromide 0.1 mg/kg for muscle relaxation, followed by a continuous infusion at the rate of 0.05 mg/kg/h until the sternum closure.
  Intraoperative analgesia: fentanyl in fractions, up to the total dose of 20-30 μg/kg.
  Sevoflurane concentration in exhaled gas will be adjusted according to patient's haemodynamic parameters and the level of anaesthesia, as assessed with BIS, with a target range of 40-60.
  Other Names: Sevoflurane anaesthesia
  Arms: Sevoflurane

SUMMARY:
The purpose of the present study is to assess, by near infrared spectroscopy with INVOS oximeter during vascular occlusion test (VOT), the influence of cardiopulmonary bypass on tissue saturation in thenar muscle.

The secondary aim is to compare the effects of propofol and sevoflurane anaesthesia on tissue saturation.

It is a prospective, randomized, open-label study. Sixty cardiac surgery patients will receive either propofol or sevoflurane anaesthesia. Three-minute VOT will be performed at the following time points: 30 minutes after anaesthesia induction, directly after sternotomy, 20 and 40 minutes after aortic cross-clamping, 20 minutes after aortic cross-clamp removal, and 45 minutes after weaning of cardiopulmonary bypass (CPB).

Group and time effects on tissue saturation will be analysed with ANOVA and post hoc Tukey's test.

DETAILED DESCRIPTION:
Near-infrared spectroscopy (NIRS) is a modern technique for cardiac surgical patient monitoring. The NIRS method is based on Lambert-Beer's law, which defines the relationship between the concentration of a substance and reduction of the intensity of electro-magnetic radiation. This reduction results from photon absorption by chromatophores, including haemoglobin, myoglobin and cytochrome P1. Absorption at the given wave-length depends on the degree of chromatophore oxygenation, and hence allows for its assessment. NIRS is currently commonly used for the assessment of brain oximetry in thoracic aorta surgery and, increasingly often, in open-heart surgery. Algorithms for sustaining adequate brain saturation were reported to decrease the incidence of neurological complications following cardiac surgery. In recent years, NIRS was proposed as a tool for the assessment of muscle saturation under short-term ischaemia and reperfusion, referred to as the vascular occlusion test (VOT). VOT is a provocative test in which tissue saturation (StO2) is measured at a peripheral site, such as the thenar eminence, while blood flow is transiently occluded with sphygmomanometer. After reaching a predefined ischaemia time or minimal StO2 threshold, the sphygmomanometer tourniquet is rapidly deflated and blood flow in the muscle is restored. Tissue saturation measurement during VOT can identify early disturbances in tissue metabolism and perfusion. The speed of the decrease in tissue saturation on ischaemia was proposed to reflect the local metabolic rate, while the lowest tissue saturation was proposed to reflect the extent of ischaemia. The speed of tissue saturation recovery on reperfusion in shock patients was proposed as a measure of microvascular capacity to increase blood flow after transient ischaemia. The results of recent studies indicated that the speed of the fall of muscle saturation during VOT is reduced in septic shock, while a decreased speed of saturation recovery on reperfusion is related to disturbed microcirculation, for example in hypovolemic shock. An understanding of anaesthetics and of the influence of cardiac surgical procedures on tissue saturation profile during VOT is essential for the future use of this tool for the assessment of the condition of patients during CPB cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* adult
* scheduled for elective, open-heart cardiac surgical operation with use of cardiopulmonary bypass.
* signed written consent

Exclusion Criteria:

* surgeon's intention to use the radial artery for arterial bypass
* symptoms of peripheral atherosclerosis
* paresis of a limb
* autoimmune disease
* other factors that could potentially affect blood flow in the upper extremities

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2012-03; Primary Completion 2013-04 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Changes in thenar muscle saturation | During VOT performed at 6 timepoints
  Thenar muscle tissue saturation was continuously monitored using an INVOS NIRS monitor (INVOS-YM 5100C Cerebral Somatic Oximeter, Covidien, Mansfield, USA).
  Thenar muscle saturation was measured during VOT 30 minutes after anaesthesia induction, which will be regarded baseline value.
  At five another timepoints VOT was performed and changes in thenar muscle saturation were measured:
  1. directly after the sternotomy,
  2. during CPB - 20 minutes after aortic cross-clamping,
  3. 40 minutes after aortic cross-clamping,
  4. 20 minutes after the release of the aortic cross-clamp,
  5. 45 minutes after weaning of CPB.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Biedrzycka, M.D., Ph.D., Principal Investigator — Medical University of Gdańsk, Department of Cardiac Anesthesiology
Locations (1):
- Medical University of Gdańsk, Department of Cardiac Anesthesiology, Gdansk, Pomeranian Voivodeship, Poland

REFERENCES:
- [Derived] Biedrzycka A, Kowalik M, Pawlaczyk R, Jagielak D, Swietlik D, Szymanowicz W, Lango R. Aortic cross-clamping phase of cardiopulmonary bypass is related to decreased microvascular reactivity after short-term ischaemia of the thenar muscle both under intravenous and volatile anaesthesia: a randomized trial. Interact Cardiovasc Thorac Surg. 2016 Nov;23(5):770-778. doi: 10.1093/icvts/ivw232. Epub 2016 Jul 8. PMID 27401083